CLINICAL TRIAL: NCT06065449
Title: A Phase III Randomized Trial Comparing Stereotactic Body Radiation Therapy (SBRT) vs Conventional Palliative Radiation Therapy for Painful Bone Metastases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0776; NCI-2023-07923 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-09-26; First posted 2023-10-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Bone Metastases
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Standard Dose (Experimental): Participants will receive either 1 radiation treatment a day for 3 days in a row (not counting weekends or holidays), or Participants will receive 1 radiation treatment given on 1 day.
  Interventions: Drug: Radiation Therapy
- Arm 2 - High Dose (Experimental): Participants will receive either 1 radiation treatment a day for 5 days, or 1 radiation treatment given on 1 day.
  Interventions: Drug: Radiation Therapy

INTERVENTIONS:
Drug: Radiation Therapy — Arm 1: standard 8 Gy delivered in a single fraction or 20 Gy delivered in 5 fractions
  Arm 2: 16 Gy delivered in a single fraction or 27 Gy delivered in 3 fractions prescribed to planning target volume (PTV).

SUMMARY:
To compare increasing doses and different treatment schedules of stereotactic body radiation therapy (SBRT) against standard treatment scheduling.

DETAILED DESCRIPTION:
Primary Objectives:

• Pain response will be assessed at 2 weeks, 1 month, 3 months and then every 3 months post-treatment and will be determined based on International Pain Consensus Criteria between the two treatment arms. The 3-month pain response will be used as the primary endpoint in trial design and for powering the test of the study's primary hypothesis of pain response.

Secondary Objectives:

* The local failure rate will be determined by radiographic response after radiation therapy. If the radiographic reports are indeterminate, the local failure rate will be based on second consecutive radiographic report showing local progression.
* To evaluate narcotics utilization converted to OMED (oral Morphine Equivalent Dose) compared to baseline prior to radiotherapy in both treatment arms.
* To evaluate rate of re-irradiation in both treatment arms.
* To evaluate rate of pathologic fracture in both treatment arms.
* To report overall survival, time from end of radiation treatment to date of death from any cause.
* To report both acute and long-term toxicity associated with radiotherapy in both treatment arms.
* To report of rate of salvage surgery after radiotherapy in both treatment arms.
* To report quality of life outcome measures defined in PROMIS study

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologic diagnosis of solid primary malignancy with any radiographic report of bone metastases including but not limited to plain x-ray, bone scan, CT scan, MRI, PET/CT scan, PSMA scan, PET fluciclovine scan. The exception is patients diagnosed with multiple myeloma are eligible.
* Patients with any pain or discomfort at proposed treatment site.
* Patients with life expectancy of 3 months or greater.
* Patients able to complete pain assessment and quality of life surveys.
* Patients with multiple osseous sites are eligible; however, should not treat more than three separate isocenters concurrently. Additional isocenters can be treated sequentially.
* Patients with prior surgery for osseous metastases are eligible.
* Patients age 18 years or older. Pediatric patients are usually enrolled on pediatric protocols. There are no adverse data available for patients < 18 years of age treated with SBRT, therefore children are excluded from this study.
* Patients may receive systemic therapy including chemotherapy, targeted therapy, immunotherapy, or other systemic agents up to and during radiation at treating physician's discretion per standard of care.
* Patients must have adequate organ and marrow function as defined below:

platelets ≥ 40,000/mcL

* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* The effects of radiation therapy on the developing human fetus are unknown. For this reason and because radiation therapy as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

  1. Postmenopausal (no menses in greater than or equal to 12 consecutive months)
  2. History of hysterectomy or bilateral salpingo-oophorectomy.
  3. Ovarian Failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy)
  4. History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 2 weeks after completion of radiation therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with prior radiation therapy to the proposed treatment site.
* Patient with current, un-treated cord compression at treatment site.
* Patients with a radiographic or pathologic fracture at the proposed treatment site that is not mechanically stable. If this is stabilized mechanically or seen by orthopedic surgery, this site is eligible for enrollment and treated on protocol
* Patients with metastases to hand and feet.
* Patients with previously treated with radioactive isotope (e.g. Sr 89) within 30 days of randomization. This can have concomitant effects with radiation therapy.
* Patients with spinal metastases along cervical, thoracic, or lumbar spine are not eligible. However, if the primary site invades the paraspinal or spine region, these are eligible.
* Pregnant patients are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2027-06-27 (Estimated); Study Completion 2027-06-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion: an average of 1year

CONTACTS AND LOCATIONS:
Overall Officials: Quynh Nguyen, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT06065449/ICF_000.pdf